CLINICAL TRIAL: NCT00751400
Title: An Open Label, Actual Use Study in Consumers Taking an Extended-Release Over the Counter NSAID in a Naturalistic Setting
Brief Title: Naproxen Sodium Extended-Release Actual Use Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Pegus Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 13129; 2014-005268-13 (EudraCT Number)
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: Non-prescription
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naproxen Sodium ER (BAYH6689) (Experimental): subjects take one tablet Naproxen Sodium ER (extended release) every 24 hours while symptoms last for no more than 10 consecutive days for pain and no more than 3 consecutive days for fever
  Interventions: Drug: Naproxen Sodium ER (BAYH6689)

INTERVENTIONS:
Drug: Naproxen Sodium ER (BAYH6689) — Consumer use of Extended Release Naproxen Sodium

SUMMARY:
The purpose of this Study is to assess how subjects will use the investigational product in an uncontrolled, naturalistic environment.

DETAILED DESCRIPTION:
Issues on adverse event data are addressed in the Adverse Event section.

The following acronyms and abbreviations were used in the results section.

- General Educational Development (GED)

ELIGIBILITY:
Inclusion Criteria:

* Self report use of Over The Counter (OTC) analgesics
* Able to read and understand English
* Provide written informed consent (subjects 12- 17 years of age provide written as sent and/ or parent or legal guardian provide written consent)
* Purchase the investigational product

Exclusion Criteria:

* Have participated in a study involving OTC analgesics in the last 12 months
* They or someone else in the household work for a market research company, an advertising agency, a public relations firm, pharmaceutical company, as a healthcare professional, or as part of a health care practice
* Have a history of known allergies to nonsteroidal anti-inflammatory drugs (NSAIDs) (i.e., Naproxen, Ibuprofen, etc) or Aspirin
* Have a history of heart surgery in the last 60 days or plans for heart surgery in the next 60 days
* (Female subjects) are pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (23):
- United States (23):
  - Anaheim, California
  - Oceanside, California
  - San Dimas, California
  - Overland Park, Kansas
  - Anoka, Minnesota
  - Blaine, Minnesota
  - Elk River, Minnesota
  - Saint Francis, Minnesota
  - Saint Louis Park, Minnesota
  - Belton, Missouri
  - Saint Joseph, Missouri
  - Savannah, Missouri
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - Syracuse, Utah
  - West Jordan, Utah
  - Kenmore, Washington
  - Seattle, Washington
  - Snohomish, Washington

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study was conducted using newspaper ads, direct mailing, in-store pharmacy posters, and flyers. Potential subjects who learned about the study through local advertising were directed to call a toll-free number (call center at the CRO (Contract Research Organization)) where minimal screening questions were asked.
Pre-assignment Details: Once at the pharmacy, if the screening criteria were met, subjects were given an (empty) OTC (Over The Counter) package and were allowed as much time as needed to review the label. They were then told the cost of the investigational product and asked if they would like to purchase it for their own use.
Period: Overall Study
Arm/Group | Naproxen Sodium ER (BAYH6689)
Started | 497
Subjects Provided Drug | 497
Subjects Consumed Drug | 485
Subjects Provided Detailed Use Data | 467
Completed | 487
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292
  Male | 205
Education [Number; unit: participants]
  8th grade or less | 6
  Some high school | 21
  High school graduate, GED, or certificate | 119
  Some college or technical school | 185
  College graduate | 117
  Post-graduate degree | 49
  Missing | 0
Literacy [Number; unit: participants] — Rapid Estimate of Adult Literacy in Medicine (REALM) scores range from 0-66 (single scale): a score of 61 or greater is considered normal literacy; a score of 60 or less is considered low literacy.
  participants
    Normal | 437
    Low | 56
    No REALM Score | 4
Prior Analgesic Use [Number; unit: participants] — Heavy analgesic user: 30 or more doses of Over The Counter (OTC) analgesics per month (self reported based on categorical responses). Regular analgesic user: 5 to 29 doses of OTC analgesics per month (self reported based on categorical responses).
  participants
    Heavy | 148
    Regular | 349
Race [Number; unit: participants]
  White | 399
  Black | 56
  Hispanic | 3
  Asian | 8
  Other | 31
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Use Days With One or More Misuse Occasions
Description: Misuse occasion: any reported use of 2 or more tablets within a 22 hour period (included use of 2 tablets in 1 dose or the use of 1 tablet at one time and 1+ tablets at a later time within the same 22 hour period). Use-days were calculated based on days in which there was subject-reported product consumption, meaning that if a tablet was consumed on a day this resulted in 1 use-day. If a subject reported product consumption on 3 different days this resulted in 3 use-days. The cumulative expression of use-days is the total number of use-days reported by all subjects with follow up data.
Time Frame: 1 month
Population: Number of subjects reflects subjects that completed at least one interview and provided use information for the previous 5 days
Measure: Number; unit: days
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
days
  use days without a misuse occasion | 2112
  use days with a misuse occasion | 294

2. Secondary Outcome: Dosing Occasions With One and More Than One Tablet Taken
Description: Dosing occasion means a single occasion in which a subject reported consuming the study drug. Multiple dosing occasions were possible throughout one use-day. For example, if a subject took one tablet at 6 am this would result in one dosing occasion. If the same subject took one tablet later that same day at 8 pm this would result in a second dosing occasion.
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: dosing occasions
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
dosing occasions
  only one tablet taken | 2500
  more than one tablet taken | 66

3. Secondary Outcome: Use Days With and Without Next Dose Less Than 22 Hours Later
Description: Use-days were calculated based on days in which there was subject-reported product consumption, meaning that if a tablet was consumed on a day this resulted in one use-day. If a subject reported product consumption on three different days this resulted in three use-days. The cumulative expression of use-days is the total number of use-days reported by all subjects with follow up data.
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: days
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
days
  no dose less than 22 hours later | 2175
  at least one dose less than 22 hours later | 231

4. Secondary Outcome: Number of Subjects With and Without More Than One Tablet Taken Per Dose
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
participants
  never took more than one tablet per dose | 440
  took more than one tablet per dose | 27

5. Secondary Outcome: Number of Subjects With and Without Next Dose Less Than 22 Hours Later
Description: This Outcome is a measure of subjects while Outcome Measure 3 provides the outcome as a measure of cumulative number of use-days for all subjects involved.
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
participants
  no doses less than 22 hours later | 359
  at least one dose less than 22 hours later | 108

6. Secondary Outcome: Number of Subjects With and Without More Than 660 mg at Least Once
Description: This measure refers to number of subjects that exceeded 660 mg of naproxen sodium per day at least once during the reporting period. The maximum dose (660 mg) may have been exceeded with one dose (if a subject consumed two tablets in one dosing occasion) or may have been exceeded throughout the course of a use-day (if a subject took one tablet in one dosing occasion and then later in the same day took one or more tablets in another dosing occasion).
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
participants
  not more than 660 mg | 344
  more than 660 mg at least once | 123

7. Secondary Outcome: Average Daily Dose
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
mg | 722 (233.4)

8. Secondary Outcome: Number of Subjects That Have Taken Study Drug on More Than 10 Consecutive Days and Not on More Than 10 Consecutive Days
Description: This measure is reporting how many subjects exceeded the label limit for consecutive days of study drug dosing
Time Frame: 1 month
Population: number of subjects reporting at least one tablet taken at any point during study
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 485
participants
  not more than 10 consecutive days | 376
  more than 10 consecutive days | 109

9. Secondary Outcome: Number of Total Dosing Occasions Per Subject
Description: as for outcome 2
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dosing occasions
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
dosing occasions | 5.5 (3.7)

10. Secondary Outcome: Number of Dosing Occasions Per Subject That Exceeded 660 mg
Description: as for outcome 2
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dosing occasions
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 467
dosing occasions | 0.6 (1.6)

ADVERSE EVENTS:
Arm/Group | Naproxen Sodium ER (BAYH6689)
Serious Adverse Events (participants affected / at risk) | 3/485
Other Adverse Events (participants affected / at risk) | 111/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=485)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=485)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Dental discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 10 (12)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Sluggishness (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood iron decreased (Investigations) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 10 (10)
Migraine (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No control group, detailed data collected for up to 10 days during 1 month followup, data recall by subjects may vary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less